CLINICAL TRIAL: NCT03385031
Title: Prospective Validation of 3D Dose Metrics as Selection Criteria for Adaptive Radiotherapy in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: P0268
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Dose-guided radiation therapy; CBCT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: whole breast irradiation, CBCT imaging at first and last fraction of radiotherapy treatment
  Interventions: Other: CBCT imaging
- group 2: simultaneous integrated boost, CBCT imaging at first and last fraction of radiotherapy treatment
  Interventions: Other: CBCT imaging
- group 3: patients with seroma at start radiation treatment (whole breast irradiation or simultaneous integrated boost), CBCT imaging at first and last fraction of radiotherapy treatment
  Interventions: Other: CBCT imaging

INTERVENTIONS:
Other: CBCT imaging — CBCT imaging at first and last fraction of radiotherapy treatment

SUMMARY:
In a retrospective study the investigators defined quantitative action levels based on dose and volume measures for adaptive radiation therapy in breast cancer patients (Zegers et al. Acta Oncol 2017). The aim of this study is to validate these parameters in a prospective study.

DETAILED DESCRIPTION:
During radiotherapy, changes in patient anatomy or positioning can result into differences in dose deposition, which is the main factor influencing tumor control or side-effects. Dose-guided radiation therapy is the systematic evaluation of the dose delivery during treatment for an individual patient with the aim to adapt the treatment if needed. Recalculation of the dose during treatment can be performed using the imaging information during treatment. In a retrospective study the investigators defined quantitative action levels based on dose and volume measures for adaptive radiation therapy in breast cancer patients (Zegers et al. Acta Oncol 2017). The aim of this study is to validate these parameters in a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients
* Planned for external beam radiation treatment.
* Whole breast irradiation or Simultaneous integrated boost

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: 1. Whole breast irradiation (N=10)
  2. Simultaneous integrated boost (N=10)
  3. Patients with seroma at start radiation treatment (N=10)
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Validation of quantitative action levels | 3-4 weeks (time between 1st and last fraction of radiotherapy)
  Evaluation of DVH parameters on the CBCT of the 1st and last fraction of radiotherapy treatment. Evaluate if the changes during treatment are within the thresholds set by the previous retrospective study; are parameters within predefined criteria yes/no

SECONDARY OUTCOMES:
Automatic re-delineation | 3-4 weeks (time between 1st and last fraction or radiotherapy)
  Evaluation of automatic re-delineation of the target volume against manual re-delineation by a radiotherapy oncologist on the CBCT of the 1st and last fraction of radiotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Karolien Verhoeven, PHD, Principal Investigator — Radiation Oncologist
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Netherlands

REFERENCES:
- [Background] Zegers CML, Baeza JA, van Elmpt W, Murrer LHP, Verhoeven K, Boersma L, Verhaegen F, Nijsten SMJJG. Three-dimensional dose evaluation in breast cancer patients to define decision criteria for adaptive radiotherapy. Acta Oncol. 2017 Nov;56(11):1487-1494. doi: 10.1080/0284186X.2017.1349334. Epub 2017 Aug 29. PMID 28849731
- See also: Three-dimensional dose evaluation in breast cancer patients to define decision criteria for adaptive radiotherapy. — https://www.ncbi.nlm.nih.gov/pubmed/?term=(Zegers+et+al.+Acta+Oncol+2017)